CLINICAL TRIAL: NCT02940977
Title: Establishment and Clinical Assessment of a Prostate Cancer (PCa) Risk Model Based on the Updated Circulating Tumor Cell (CTC) Detection Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Shen Kang Hospital Development Center (Other)
Responsible Party: Principal Investigator, Jun Qi, Head of the Urology Department, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-028
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Prostatic Neoplasms; Prostatic Adenoma
Keywords: Circulating tumor cell; Epithelial to mesenchymal transition; Prostate specific antigen (PSA); Partin table
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh blood 5 ml *2
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate cancer patients: Patients diagnosed with prostate cancer, confirmed with needle biopsy, and suitable for radical prostatectomy, and have not received any treatments before.
  Interventions: Other: Blood draws

INTERVENTIONS:
Other: Blood draws — Blood draws, from peripheral veins, each time 2 tubes, each 5 ml.

SUMMARY:
1. To elucidate the role of CTC detection in the evaluation of risk level in PCa patients, and establish a mathematic model for predicting the pathological status.
2. To explore the possible subtle change in CTC condition after radical prostatectomy.

DETAILED DESCRIPTION:
1. Detect and evaluate the CTC status (a total of 3 times: 1 day before sugery, 3/12 months after surgery) for all of the PCa patients enrolled. Analyze the CTC result with PSA level, needle biopsy and radiological imaging information.
2. Analyze the difference in CTC amount/Epithelial-Mesenchymal ratio between patients in different D'Amico risk level(low/intermediate/high).
3. Establish a mathematic model based on the CTC results and pathological condition observed in operation (OC, organ confined; EPE, extraprostatic extension; SVI, seminal vesicle invasion; LNI, lymph node invasion), and compare this model with the latest version of Partin table.
4. Detect and compare the CTC and PSA level 3/12 months after surgery. Evaluate the radiological condition in 12 months after blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with PCa by biopsy, for the first time.
2. Clinical assessed suitable for radical prostatectomy
3. Age ≥ 18 years, able to provide written informed consent
4. No prior systematic or regional treatment for PCa.
5. No neuro-endocrine differentiation or small cell PCa pattern.
6. ECOG status 0-1
7. Expected life span ≥ 12 months.
8. Multiorgan function (heart, lung, liver, kidney) able to tolerate radical prostatectomy, and meet the standard of this study.

Exclusion Criteria:

1. Severe concomitant disease or infection.
2. ALT or AST > 2.5 ULN, or total bilirubin > 1.5 ULN; Creatinine >177umol/L(2.5mg/dL)；Plt < 100,000/uL, Neutrophil <1,500/uL.
3. Known or suspected brain metastasis or leptomeningeal carcinomatosis.
4. Another malignancy in the last 5 years, excluding completely cured melanoma.
5. Severe cardiovascular disease, including:

   Myocardial infarct within 6 months; Uncontrolled angina pectoris within 3 months; Congestive heart failure; Ventricular arrhythmia history with clinical significance; Morbiz type Ⅱ or complete heart block
6. Major surgery (general anesthesia) within 4 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with prostate cancer, confirmed with needle biopsy, and suitable for radical prostatectomy, and have not received any treatments before.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor cell (CTC) total number and epithelial-intermediate-mesenchymal ratio detected by CTC enrichment and FISH technique | 1 day before operation
  This step should be completed within the day when the peripheral venous blood is drawn.
Pathological findings (whether the patient has: 1.OC, organ confined; 2.EPE, extraprostatic extension; 3. SVI, seminal vesicle invasion; 4. LNI, lymph node invasion) during the radical prostectomy, confirmed by pathology section result | On the day of operation
  The pathology section evaluation will be done by two pathologists independently. A third pathology expert will join to make a final decision if opposite results are given by the two pathologists.
CTC total number and epithelial-intermediate-mesenchymal ratio detected by CTC enrichment and FISH technique | 3 months after operation
  This step should be completed within the day when the peripheral venous blood is drawn.
CTC total number and epithelial-intermediate-mesenchymal ratio detected by CTC enrichment and FISH technique | 12 months after operation
  This step should be completed within the day when the peripheral venous blood is drawn.

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) level measurement using peripheral venous blood | 3 months after operation
  The blood should be drawn together with that for CTC detection
Prostate specific antigen (PSA) level measurement using peripheral venous blood | 6 months after operation
  The blood should be drawn together with that for CTC detection
PSA level measurement using peripheral venous blood | 9 months after operation
  The blood should be drawn together with that for CTC detection
Radiological evaluation including isotope bone scanning and pelvic magnetic resonance imaging (MRI) scan | 12 months after operation
  Radiological evaluation should be conducted after the blood is drawn for CTC and PSA detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes